CLINICAL TRIAL: NCT02657954
Title: Cognitive Rehabilitation for Homeless OEF/OIF/OND Veterans
Brief Title: ASPIRE Cognitive Enhancement Study
Acronym: ACES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1972-I
Record Dates: First submitted 2015-12-17; First posted 2016-01-18 (Estimated); Results first posted 2023-12-12 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-02

CONDITIONS: Homelessness; Mental Health Conditions
Keywords: Homeless persons; Veterans; Mental disorders; Cognition; Rehabilitation
MeSH Terms: conditions — Mental Disorders | interventions — HCE

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Compensatory Cognitive Training (CCT) (Experimental): Compensatory Cognitive Training
  Interventions: Behavioral: CCT
- Holistic Cognitive Education (HCE) (Active Comparator): Holistic Cognitive Education
  Interventions: Behavioral: HCE

INTERVENTIONS:
Behavioral: CCT — 10-week Compensatory Cognitive Training
  Arms: Compensatory Cognitive Training (CCT)
Behavioral: HCE — 10-week Holistic Cognitive Education
  Arms: Holistic Cognitive Education (HCE)

SUMMARY:
Cognitive impairments are present in up to 80% of homeless individuals, and may contribute to homelessness in Operation Enduring Freedom / Operation Iraqi Freedom / Operation New Dawn (OEF/OIF/OND) Veterans. The investigators propose to investigate these issues in homeless, treatment-seeking returning Veterans, who arguably face multiple potential barriers to recovery and reintegration, and with whom there is the greatest opportunity to prevent long-term homelessness. The investigators plan to conduct a 15-week randomized controlled trial of an evidence-based, 10-week Compensatory Cognitive Training (CCT) intervention vs. an education control condition to examine the effects of cognitive rehabilitation in this Veteran population. The investigators expect CCT-associated improvements in cognition and functional skills and generalization to reduced levels of disability, along with improved community reintegration outcomes. By attending to and treating cognitive impairments, the investigators can potentially prevent future homelessness and its negative health consequences, resulting in both healthcare cost savings and improved quality of life for Veterans.

DETAILED DESCRIPTION:
This study integrates cognitive rehabilitation in residential care for homeless Veterans. In a 15-week randomized controlled trial, the investigators will compare an evidence-based, 10-week Compensatory Cognitive Training (CCT) intervention to an education control condition for homeless Veterans with cognitive impairment. CCT aims to improve real-world cognitive performance by teaching strategies to improve prospective memory (remembering to do things), attention, learning/memory, and executive functioning. Strategies to reduce stress and improve sleep are also included. CCT has been shown to improve cognition, functional capacity, neurobehavioral symptom severity, and quality of life in individuals with cognitive impairment associated with psychiatric illness and in Veterans with traumatic brain injury (TBI). During the trial, assessments will be administered at baseline, 5 weeks, 10 weeks, and 15 weeks, and monthly follow-up phone calls will assess housing and employment/education status for one year following program discharge. The investigators expect CCT-associated improvements in cognition and functional skills (co-primary outcomes) and generalization to reduced levels of disability, along with improved community reintegration outcomes (better housing stability, participation in work or school, and healthcare appointment attendance). If effective, the CCT intervention could be exported to the 80+ residential VA programs serving homeless Veterans. The investigators thus propose the following aims:

Aim 1. Investigate the efficacy of cognitive rehabilitation in homeless returning Veterans with mental health conditions and cognitive impairment by conducting a randomized controlled trial of Compensatory Cognitive Training (CCT) vs. education control for 10 weeks, with a 5-week follow-up, followed by 1 year of monthly post-discharge follow-up phone calls to assess community reintegration outcomes.

H1a: Positive CCT-associated effects on cognition, functional capacity (co-primary outcomes), and disability will emerge over the 15-week study.

H1b: Positive CCT-associated effects on community reintegration outcomes (housing stability, participation in employment/education, healthcare appointment attendance) will be detected at the end of the 1-year follow-up.

Aim 2. Investigate mechanisms of CCT effects. H2: Improved cognition and cognitive strategy use will mediate improvements in functional capacity, disability, and community reintegration.

Exploratory Aim 3. Investigate moderators of CCT effects. Presence and severity of Posttraumatic Stress Disorder (PTSD), depression, history of substance abuse, and TBI, as well as duration of homelessness and baseline cognitive functioning, will be explored as potential moderators of CCT effects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Any race/ethnicity
* Age 18-55
* Receiving residential treatment at the VA San Diego Aspire Center
* Meets criteria for Aspire Center program entry

  * OEF/OIF/OND Veteran
  * Presence of at least one DSM-V mental health condition
  * Does not meet criteria for substance use disorder for 28 days prior to admission
  * Homeless or unstably housed
  * Not a sex offender or violent offender
  * Capable of performing activities of daily living and transfers
  * Not judged by a clinician to be at current risk to self or others
* Has cognitive impairment in at least one cognitive domain (i.e., T-score <40)
* Able to speak and read English
* Capable of and willing to provide signed informed consent

Exclusion Criteria:

None.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth W. Twamley, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keller AV, Muller-Cohn CM, Austin TA, Jak AJ, Twamley EW. Neuropsychological functioning, neurobehavioral symptoms, and community reintegration in unstably housed veterans with mental health conditions. Clin Neuropsychol. 2023 Nov;37(8):1728-1744. doi: 10.1080/13854046.2023.2176364. Epub 2023 Feb 11. PMID 36772819

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 79 participants were enrolled and randomized to a condition and were included in intent to treat analyses, but 10 dropped out before starting their assigned intervention (5 in each arm).
Period: Overall Study
Arm/Group | Compensatory Cognitive Training (CCT) | Holistic Cognitive Education (HCE)
Started | 39 | 40
Received at Least One Session | 34 | 35
Completed | 20 | 26
Not Completed | 19 | 14

BASELINE CHARACTERISTICS:
Population: 79 participants enrolled and baseline tested; 10 did not receive intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Compensatory Cognitive Training (CCT) | Holistic Cognitive Education (HCE) | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (7.7) | 37.0 (6.9) | 37.3 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 39 | 39 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 12 | 21
  Not Hispanic or Latino | 30 | 28 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 5 | 9
  White | 29 | 25 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Deficit Score From Expanded MATRICS Consensus Cognitive Battery (MCCB)
Description: Global Deficit Score (composite score) from MATRICS Consensus Cognitive Battery plus Delis-Kaplan Executive Function System (D-KEFS) subtests (Verbal Fluency, Color-Word Interference), Trail Making Test, Part B
  Global deficit score range = 0-5, lower scores are better, higher scores are worse. For change in global deficit score, higher is better.
Time Frame: baseline to 15 weeks
Population: All participants who completed a baseline assessment (i.e., intent to treat sample)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compensatory Cognitive Training (CCT) | Holistic Cognitive Education (HCE)
Number analyzed (Participants) | 39 | 40
score on a scale | 0.26 (0.47) | .14 (.12)

2. Primary Outcome: Change in UCSD Performance-Based Skills Assessment-Brief (UPSA-B)
Description: Performance-based functional capacity in finance and communication
  UPSA scores range from 0-100, higher scores are better. For change in UPSA scores, higher is also better.
Time Frame: baseline to 15 weeks
Population: All participants with baseline data included (i.e., intent to treat sample)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compensatory Cognitive Training (CCT) | Holistic Cognitive Education (HCE)
Number analyzed (Participants) | 39 | 40
score on a scale | 8.3 (8.9) | 8.3 (8.6)

3. Secondary Outcome: Change in World Health Organization Disability Assessment Schedule (WHODAS) 2.0
Description: Measure of level of disability
  WHODAS scores range from 0-100, higher scores are worse. For change in WHODAS scores, higher scores are also worse.
Time Frame: baseline to 15 weeks
Population: All participants with baseline data (i.e., intent to treat sample)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compensatory Cognitive Training (CCT) | Holistic Cognitive Education (HCE)
Number analyzed (Participants) | 39 | 40
score on a scale | -5.6 (13.2) | -4.5 (8.4)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from baseline assessment to 12-months post-discharge. Study length was variable due to variability in time of treatment center discharge (study length was 1.5 years on average).
Arm/Group | Compensatory Cognitive Training (CCT) | Holistic Cognitive Education (HCE)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 0/39 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT02657954/Prot_SAP_000.pdf